CLINICAL TRIAL: NCT00447486
Title: A Multicentre, Randomised, Double-Blind, Placebo and Naproxen (500mg) BID Controlled, Phase II Proof of Concept, Parallel Group Study to Assess the Efficacy and Safety of Oral GW842166 at Two Dose Levels Administered for 4 Weeks in Adults With Osteoarthritis of the Knee
Brief Title: A Study of GW842166 in Adults With Osteoarthritis Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CBA109389
Record Dates: First submitted 2007-03-12; First posted 2007-03-14 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2009-05

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis,; knee,; GW842166,; pain,; efficacy,; safety
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain

INTERVENTIONS:
Drug: GW842166

SUMMARY:
The purpose of this study is to determine whether GW842166 is effective in the treatment of osteoarthritis pain of the knee.

ELIGIBILITY:
Inclusion Criteria:

* male or female outpatient, >= 40 years of age
* meets ACR clinical and radiographic criteria for classification of idiopathic (primary) osteoarthritis of the knee with symptom duration for at least 3 months
* meets ARA functional status requirements
* meets WOMAC pain subscale score requirements
* has taken analgesics for the treatment of their knee OA for at least 4 out of 7 days in each of the 4 weeks preceding screen

Exclusion Criteria:

* any pre-specified clinical/biological/ECG abnormality
* any pre-specified drug sensitivity
* history of peptic ulceration or GI bleeding
* use of protocol-specified medications
* secondary cause of knee OA
* lower extremity surgery within 6 months of screening
* use of analgesics other than allowed per protocol
* use of corticosteroids or hyaluronan outside of allowed window prior to screening

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2007-04

PRIMARY OUTCOMES:
The pain subscale score on the Western Ontario and McMasters Universities OA Index (WOMAC) taken at Day 28 compared to baseline | 4 Weeks

SECONDARY OUTCOMES:
WOMAC pain subscale, stiffness, physical function scores and patient and physician global assessments | 4 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, BSc MB PhD, Study Director — GlaxoSmithKline
Locations (19):
- Denmark (2):
  - GSK Investigational Site, Hvidovre
  - GSK Investigational Site, Odense C
- Germany (7):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Schmiedeberg, Saxony
  - GSK Investigational Site, Berlin, State of Berlin
- Spain (5):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Centelles
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Petrer/Alicante
  - GSK Investigational Site, Santiago de Compostela
- Sweden (5):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Helsingborg
  - GSK Investigational Site, Höllviken
  - GSK Investigational Site, Stocholm
  - GSK Investigational Site, Upplands Vasby